CLINICAL TRIAL: NCT05886140
Title: Carrellizumab Combined With Albumin-binding Paclitaxel in the Treatment of Locally Late Stage or Relapsed Metastatic Cutaneous Squamous Cell Carcinoma: a Single-arm, Open, Multicenter, Prospective Clinical Study
Brief Title: Carrilizumab Combined With White Purple for Squamous Cell Carcinoma of Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhang Peng, Deputy chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-SHR-1210-cSCC-002
Record Dates: First submitted 2023-05-14; First posted 2023-06-02 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-05

CONDITIONS: Squamous Cell Carcinoma of the Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carrilizumab with albumin-binding paclitaxel (Experimental): All enrolled patients received carrilizumab combined with albumin-binding paclitaxel.
  Interventions: Drug: Carrilizumab with albumin-binding paclitaxel

INTERVENTIONS:
Drug: Carrilizumab with albumin-binding paclitaxel — All enrolled patients received carrilizumab combined with albumin-binding paclitaxel.

SUMMARY:
This study intends to conduct a single-arm, prospective and open clinical study, using carrellizumab combined with albumin-binding paclitaxel regimen for first-line treatment of squamous cell carcinoma of the skin, including 24 patients with squamous cell carcinoma of the skin, to further confirm the efficacy and safety of Carrellizumab combined with albumin-binding paclitaxel in the treatment of squamous cell carcinoma of the skin.

DETAILED DESCRIPTION:
This study intends to conduct a single-arm, prospective and open clinical study in the Department of Bone and Soft Tissue of Henan Cancer Hospital. The first-line treatment of squamous cell carcinoma of the skin with carrellizumab combined with albumin-binding paclitaxel regimen is adopted. 24 patients with squamous cell carcinoma of the skin are included. It is intended to further confirm the efficacy and safety of carrellizumab combined with albumin-binding paclitaxel in the treatment of cutaneous squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥18 years old; ECOG score 0~1, organ function is good; Histologically confirmed first-line treatment for locally advanced or relapsed metastatic squamous cell carcinoma of the skin.

There were measurable tumor lesions evaluated by MRI or CT during the 21 days prior to enrollment;

If you have received antitumor therapy, the following conditions should be met:

1. The interval between systemic radiotherapy and the first dose in this study was ≥3 weeks, and the interval between local radiotherapy was ≥2 weeks;
2. The interval between previous chemotherapy, targeted therapy, biotherapy, endocrine therapy and other antitumor therapies and the first administration in this study was ≥4 weeks; Normal function of major organs (within 14 days prior to treatment); For female patients who are not menopausal or have not been surgically sterilized: consent to abstinence from sex or use of effective contraceptive methods during treatment and for at least 7 months after the last dose in the study treatment; The patients voluntarily participated in this study and signed the informed consent.

Who can be included as judged by the researcher.

Exclusion Criteria:

Previously received anti-PD-1, anti-PD-L1, anti-PD-L2 drug therapy; Also receiving antitumor therapy in other clinical trials; Had major surgical operations within 4 weeks prior to enrollment, or had not fully recovered from such operations; Serious heart disease or discomfort or concomitant disease that, according to the judgment of the investigator, seriously endangers the safety of the patient or affects the completion of the study; Allergic reactions: Patients who are allergic to the investigational drug or to any investigational drug component in the chemotherapy regimen are not recommended for inclusion.

Pregnant and lactating women, fertile women who tested positive for baseline pregnancy tests, or patients of childbearing age who did not want to take effective contraceptive measures during the entire trial period and within 6 months after the last study; Those considered unsuitable for inclusion by researchers.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | It is estimated to take about 60 months from the start of enrollment to the end of the experiment.
  The proportion of tumor volume reduction that reaches the predetermined value and maintains the minimum time limit.

SECONDARY OUTCOMES:
Progression-Free-Surviva | The estimated time from enrollment to disease progression is about 24 months.
  The time from the start of treatment to the appearance of secondary growth

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No